CLINICAL TRIAL: NCT02703584
Title: Co Administration of GnRH Agonist and hCG for Final Oocyte Maturation- A Randomized Controlled Trial
Brief Title: Co Administration of GnRH Agonist and hCG for Final Oocyte Maturation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03012016
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2016-06

CONDITIONS: Infertility
Keywords: Double trigger
MeSH Terms: conditions — Infertility | interventions — Buserelin; Saline Solution; Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double trigger (Experimental): Triggering of ovulation with GnRH agonist ( Suprefact 0.5mg) + hCG ( Pregnyl 10,000IU)
  Interventions: Drug: Buseralin; Drug: pregnyl
- control (Placebo Comparator): Triggering of ovulation with hCH ( Pregnyl 10,000IU) + Placebo
  Interventions: Other: Placebo; Drug: pregnyl

INTERVENTIONS:
Drug: Buseralin
  Other Names: Suprefact
  Arms: Double trigger
Other: Placebo
  Other Names: normal saline
  Arms: control
Drug: pregnyl
  Other Names: hCG

SUMMARY:
All the studies, demonstrating improved oocyte maturity and high pregnancy rate with the dual trigger are all retrospective. The investigators therefore aim to perform a prospective randomized controlled study in normal responders, comparing cycles triggered with hCG to those triggered with hCG+GnRH agonist.

DETAILED DESCRIPTION:
A prospective, randomized, double blinded clinical trial. Patients will undergo standard clinical and hormonal investigation as usual for IVF. Patients that will be given the standard GnRH antagonist IVF protocol will be prospectively randomized into two groups: 1. hCG group- will be triggered for final follicular maturation with hCG (Pregnyl 10,000IU) as is usual and placebo (normal saline) - 36 hours prior to oocyte aspiration. 2. The Double trigger group- will receive GnRH agonist (Suprefact 0.5 mg) and hCG (Pregnyl 10,000IU) 36 hours prior to the oocyte aspiration. All patients will be supplemented with the usual progesterone preparation (vaginal progesterone suppositories) for luteal support.

In order to increase the rate of MII from to 65% to 80% with an alpha error of 5% and beta error of 80% the sample size needed is 276 total patients in both groups or 138 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* Women during one of their first 3 IVF cycle attempts
* Women between the ages of 18-42.
* BMI (body mass index) of 18-35.
* AMH (Anti mullerian hormone) > 1 ng/ml
* FSH˂ 20 IU/L.
* Informed consent.

Exclusion Criteria:

* Women with low ovarian response
* Previous enrollment in this study.
* AFC>20
* E2 above 15,000 pmol/l at the trigger day.
* hypersensitive to Suprefact/Pregny/gonal F/Purigon/Menopur/progesterone, and/or their ingredients/components of the formulation
* primary ovarian failure
* pregnancy and breast-feeding
* active blood clots
* undiagnosed uterine or genital bleeding
* endometriosis
* uncontrolled hypertension;
* uncontrolled diabetes
* abnormal liver and kidney functions
* abnormal ECG, e.g. QT prolongation and torsades de pointes
* cancers/tumors, e.g. pituitary adenomas, ovarian cysts, etc.
* HIV, HBV and HCV infections
* low bone mineral density (BMD) and an increased risk of bone fracture, such as chronic alcohol and/or tobacco use, presumed or strong family history of osteoporosis or chronic use of drugs that can reduce bone mass such as anticonvulsants or corticosteroids
* suicidal tendency, history or disposition to seizures, state of confusion, clinically relevant psychiatric disorders, and brain lesions
* Use of an investigational drug or participation in an investigational study within 30 days prior to this study.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes | 2 days after randomization
  We will gather the information regarding the number of mature oocytes 2 days after the triggering- ( randomization)

SECONDARY OUTCOMES:
Blastocyst rate | 8 days after the randomization

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Casper, MD, Principal Investigator — Scientific Director TRIO IVF
Locations (1):
- TRIO Fertility, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozelci R, Yenigul NN, Dilbaz S, Dilbaz B, Aldemir O, Kaplanoglu I, Gucel F, Baser E, Tekin OM. The Association of ICSI Outcomes with Semen and Blood Bisphenol A Concentrations of the Male Partner. Reprod Sci. 2024 May;31(5):1323-1331. doi: 10.1007/s43032-023-01446-y. Epub 2024 Jan 11. PMID 38212582
- [Derived] Haas J, Bassil R, Samara N, Zilberberg E, Mehta C, Orvieto R, Casper RF. GnRH agonist and hCG (dual trigger) versus hCG trigger for final follicular maturation: a double-blinded, randomized controlled study. Hum Reprod. 2020 Jul 1;35(7):1648-1654. doi: 10.1093/humrep/deaa107. PMID 32563188